CLINICAL TRIAL: NCT05360134
Title: Efficacy and Safety of Platelet Augmentation Using Carica Papaya Leaf Extract in Live Donor Liver Transplantation Recipients - a Pilot Randomized Controlled Trial
Brief Title: Platelet Augmentation Using C. Papaya Leaf Extract in Live Donor Liver Transplantation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Institute of Liver and Biliary Sciences, India (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ILBS-LDLT-01
Record Dates: First submitted 2022-04-25; First posted 2022-05-04 (Actual); Last update posted 2022-05-04 (Actual); Status verified 2022-04

CONDITIONS: Thrombocytopenia
MeSH Terms: conditions — Thrombocytopenia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Carica Papaya Arm (Experimental): 1100mg of Carica Papaya Leaf extract administered three times daily for upto one week preoperatively and from post-operative day 3 to day 7.
  Interventions: Drug: Carica Papaya Leaf Extract
- Placebo Arm (Placebo Comparator): Placebo administered 3 time daily for upto one week preoperatively and from post-operative day 3 to day 7.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Carica Papaya Leaf Extract — Carica Papaya Leaf Extract 1100 mg X TDS started at least 3 days preoperatively and continued on post operative day 3 to day 7
  Arms: Carica Papaya Arm
Other: Placebo — Placebo will be given in a similar manner
  Arms: Placebo Arm

SUMMARY:
This project is a pilot randomized controlled trial aimed at investigating the potential of Carica Papaya Leaf Extract, available in a marketed pill formulation, in increasing platelet counts in live donor liver transplant recipients. Carica Papaya leaf extract has shown positive results in increasing platelet counts in various medical conditions such as Dengue, Immune thrombocytopenic purpura and chemotherapy induced thrombocytopenia. Thrombocytopenia i.e. low platelet counts are a common occurrence in patients with chronic liver disease undergoing live donor liver transplant. It has been observed in previous studies that live donor liver transplant recipients who have persistent thrombocytopenia have significantly worse outcomes as compared to patients who have higher platelet counts. Positive results in this study lead to further studies in assessing the impact of platelet augmentation in live donor liver transplant recipients.

ELIGIBILITY:
Inclusion Criteria:

* All consenting adults who are planned to undergo live donor liver transplant with platelet counts less than or equal to 75000/μL preoperatively.

Exclusion Criteria:

* Patients who do not consent
* ALF & ACLF
* Pediatric transplant recipients
* Allergic to papaya
* Preoperative platelet counts >75,000/ μL
* Recent history of DVT

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2022-10-01 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
POD 7 Platelet Counts | 7th post-operative day

SECONDARY OUTCOMES:
Pre-operative platelet counts | 1 day prior to surgery
Intra-operative blood loss and transfusion requirements | Day 0
Incidence of Early allograft dysfunction | First 7 days following live donor liver transplant
Incidence of prolonged post-operative drainage | First 14 days following live donor liver transplant

CONTACTS AND LOCATIONS:
Overall Officials: Viniyendra Pamecha, FEBS, Study Director — Institute of Liver & Biliary Sciences
Locations (1):
- Institute of Liver & Biliary Sciences, New Delhi, National Capital Territory of Delhi, India

IPD SHARING:
Plan to Share IPD: No